CLINICAL TRIAL: NCT07140276
Title: An Integrated Substance Abuse-Domestic Violence (SADV) Treatment Outcome Study: A Stage 1 Trial for SADV
Brief Title: An Integrated Substance Abuse-Domestic Violence (SADV) Treatment Outcome Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10492; RDA018284A (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Substance Abuse; Domestic Violence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Men referred by the courts or probation for treatment of substance use who have domestic violence related problems.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual SADV Therapy (Experimental): Men referred from court and probation for treatment of substance use and domestic violence related problems will receive 12 weeks of individual therapy that focuses on SADV.
  Interventions: Behavioral: Individual Therapy
- Manualized comparison condition (Experimental): Men referred from court and probation for treatment of substance use and domestic violence related problems will receive 12 weeks of therapy using the manual provided that focuses on substance use only.
  Interventions: Behavioral: Individual Drug Counseling manual

INTERVENTIONS:
Behavioral: Individual Therapy — 12 weeks individual psychotherapy
  Arms: Individual SADV Therapy
Behavioral: Individual Drug Counseling manual — 12 weeks using the manual provided
  Arms: Manualized comparison condition

SUMMARY:
Investigators will conduct a randomized trial comparing individual SADV to a manualized comparison condition that focuses on substance use only.

DETAILED DESCRIPTION:
The randomized trial will be informed by previous work developing and refining the interventions and training materials used in the randomized trial.

The focus of this registration is the randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* referred by the courts or probation for treatment of substance use and domestic violence and who
* meet current DSM-IV criteria for substance dependence (alcohol, cocaine and marijuana, and who have used that substance within the 30 days prior to the screening session)
* report physical violence in an intimate relationship (pushing, slapping, kicking) within 30 days prior to screening
* can read English at a 6th grade level.

Exclusion Criteria:

* Currently in withdrawal from substances and in need of detoxification (such individuals may be re-evaluated following detoxification)
* Have cognitive impairment (a mini mental state score <25)
* Have psychomotor epilepsy (e.g. impulsivity or rage related symptoms secondary to a seizure disorder, as this medical diagnosis is likely to be a confound in the proposed study)
* Have major medical complications such as a head injury/trauma, or HIV dementia that may also be a confound in the study interventions
* Currently receiving either substance abuse or IPV treatment elsewhere
* Have a lifetime history of any psychotic or bipolar disorder
* Currently suicidal or homicidal.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-07-03 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
Mean Days of substance use | Weekly up to 12 weeks
  Days of substance use weekly from each participant endorsed as Y/N, by Self-report using time line follow back method, verified by alcohol concentration and urine toxicology
Mean Days of physical violence use | Weekly up to 12 weeks
  Days of physical violence use weekly from each participant endorsed as Y/N, by Self-report using time line follow back method, verified by female collateral informant

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Easton, PhD, Principal Investigator — University of Rochester
Locations (1):
- Yale New Haven Health System, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No